CLINICAL TRIAL: NCT04240925
Title: Tolerability, Safety and Efficacy of Sigh During Non-invasive Mechanical Ventilation in Patients With Motor Neuron Disease- A Pilot Study
Brief Title: Tolerability, Safety and Efficacy of Sigh Breaths During NIMV in Motor Neuron Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Nilo Riva, Principal Investigator, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SIGH_01
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Motor Neuron Disease; Respiratory Failure; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Motor Neuron Disease; Respiratory Insufficiency; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard NIMV protocol with sigh breaths (Experimental)
  Interventions: Device: NIMV with sigh breaths
- Standard NIMV protocol without sigh breaths (Active Comparator)
  Interventions: Device: Standard NIMV

INTERVENTIONS:
Device: NIMV with sigh breaths — Sigh breaths: Maximal Inspiratory pressure (IPAPmax) increased of at least 25% ( ≥ 125%) with a frequency of at least 1/200 breaths. The sigh breaths will be delivered as part of the standard NIMV protocol
  Arms: Standard NIMV protocol with sigh breaths
Device: Standard NIMV — Will be treated by standard NIMV with no sigh
  Arms: Standard NIMV protocol without sigh breaths

SUMMARY:
Non-invasive mechanical ventilation (NIMV) is the recommended standard of care as initial therapy for patients with motor neuron disease (MND) with deterioration of the respiratory function.

SIGH_01 study is aimed at investigating the tolerability, safety profile and efficacy of sigh breaths during non-invasive mechanical ventilation in patients with MND in comparison to the standard ventilation support protocol.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* MND diagnosis according to El-Escorial criteria
* Non-invasive ventilation indications in accordance with the international guidelines

Exclusion Criteria:

* Inability to adhere to study visit schedule or lack of reliable caretaker
* Presence of dementia
* History of arrhythmia, heart failure or pneumothorax

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in nocturnal oxygen desaturation index (ODI) assessed by transcutaneous nocturnal oximetric registration | Evaluation will be performed before NIMV initiation and two months after

SECONDARY OUTCOMES:
Changes in the arterial blood PCo2 concentration assessed by arterial blood gas test | Evaluation will be performed before NIMV initiation and two months after
Changes in the arterial blood PO2 concentration assessed by arterial blood gas test | Evaluation will be performed before NIMV initiation and two months after
Changes in the arterial blood Ph assessed by arterial blood gas test | Evaluation will be performed before NIMV initiation and two months after
Changes in the forced vital capacity (FVC) assessed by spirometry test | Evaluation will be performed before NIMV initiation and two months after
Changes in self-perceived quality of life(QoL) assessed by 5-item Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-5). Score between 0 and 100 pts (higher score denotes worse QoL) | Evaluation will be performed before NIMV initiation and two months after
Changes in sleep quality assessed by Pittsburg Sleep Quality Index (PSQI) questionnaire. Score between 0 to 21, where higher scores denote a worse sleep quality. | Evaluation will be performed before NIMV initiation and two months after
Changes in sleep quality assessed by Numeric Rating Scale (NRS). Score between 0 to 10, where higher scores denote a worse sleep quality. | Evaluation will be performed before NIMV initiation and two months after
Changes in nocturnal dyspnoea assessed by Numeric Rating Scale (NRS). Score between 0 to 10, where higher scores denote a worse nocturnal dyspnoea. | Evaluation will be performed before NIMV initiation and two months after

CONTACTS AND LOCATIONS:
Overall Officials: nilo riva, MD,PhD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No